CLINICAL TRIAL: NCT01928017
Title: Monitoring of Thromboelastography, Platelet Function and Platelet Recovery in Haemato-oncologic Patients With Thrombocytopenia
Brief Title: Thromboelastography, Platelet Function and Platelet Recovery in Haemato-oncologic Patients With Thrombocytopenia
Status: Completed | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Elin Netland Opheim, Research fellow, University of Bergen
Other Study IDs: 2011/1881
Record Dates: First submitted 2013-08-16; First posted 2013-08-23 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Bone Marrow Diseases; Lymphoma
MeSH Terms: conditions — Bone Marrow Diseases; Lymphoma

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma specimens are kept frozen.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hematooncology patients: No intervention

SUMMARY:
This is a prospective observational clinical study to characterise abnormalities of thromboelastography (TEG) parameters in patients with chemotherapy-induced thrombocytopenia. The investigators are also studying the relationship between Multiplate analysis and bleeding in these patients and the effect of platelet transfusions on thrombopoietin level and percent reticulated platelets.

The investigators' hypothesis is that changes in TEG-parameters reflect the patients tendency to bleed.

DETAILED DESCRIPTION:
Thrombocytopenic patients are followed with blood samples (thromboelastography, Multiplate, haematology) daily, Monday to Friday for up to 30 days.

In addition bleeding evaluation is done daily ,using a standardized questionnaire. The questionnaire is filled out after interview of the patient, and som times next of kin and nurses. Nurse journals and medical journals are also used to fill in the questionnaires.

For thromboelastography (TEG) we are looking at which parameters are abnormal, and if there is other factors than platelet count that influence the results. We will also compare TEG from days with and without bleeding, to see if they differ.

For Multiplate we are doing a pilot study to see whether this analysis can be of any use at all in this group of patients. We are looking into which factors that influence the Multiplate result, and if we can see a difference in the results if the patient is bleeding.

For reticulated platelets and thrombopoietin we are studying the levels related to platelet transfusions.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for this study if:

They have a haemato-oncologic disease They have, or are expected to have, thrombocytopenia They are expected to need at least one platelet transfusion They are aged 18 years or over They consent to participate

Exclusion Criteria:

Patients are not eligible for this study if:

They have a known congenital clotting disorder They need anticoagulants regularly in the study period They have immune thrombocytopenic purpura

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital inpatients admitted to the Department of Medicine, Section for Haematology at Haukeland University Hospital will be invited to join the study if they meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
MA | 1 year
  To characterise changes in the TEG-parameter MA in patients with chemotherapy-induced thrombocytopenia

OTHER OUTCOMES:
Reticulated platelets percent | 1 year
  To investigate the effect of platelet transfusions on percent reticulated platelets.
Bleeding | 1 year
  To investigate the relationship between TEG-parameters, bleeding and need for platelet transfusion.
  To investigate the influence of HLA antibodies on risk of bleeding and transfusion complications.

CONTACTS AND LOCATIONS:
Overall Officials: Tor A Hervig, dr.med, Study Director — University of Bergen
Locations (1):
- Haukeland University Hospital, Bergen, Norway